CLINICAL TRIAL: NCT04874155
Title: A Multi-Center, Randomized, Double-Blind, Sham-Controlled Study to Evaluate the NTX100 Neuromodulation System for Patients With Medication-Refractory Primary Restless Legs Syndrome (RLS) - The RESTFUL Study
Brief Title: Noninvasive Peripheral Nerve Stimulation for Medication-Refractory Primary RLS (The RESTFUL Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noctrix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-04
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Intervention Model Description: Study consists of two phases. Phase 1: Randomized 1:1 between Active treatment and Sham control Phase 2: Non-randomized, Active treatment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Active neurostimulation (Active Comparator): Noninvasive peripheral nerve stimulation device programmed to deliver active stimulation - Phase 1
  Interventions: Device: NTX100 Neuromodulation System - Active
- Sham neurostimulation (Sham Comparator): Noninvasive peripheral nerve stimulation device programmed to deliver non-therapeutic (sham) stimulation - Phase 1
  Interventions: Device: NTX100 Neuromodulation System - Sham
- Open-Label (Active Comparator): Open-Label - Phase 2 lasting 4-wks, during which all subjects will receive open-label Active treatment
  Interventions: Device: NTX100 Neuromodulation System - Open-Label

INTERVENTIONS:
Device: NTX100 Neuromodulation System - Active — Noninvasive peripheral nerve stimulation device programmed to active mode.
  Arms: Active neurostimulation
Device: NTX100 Neuromodulation System - Sham — Noninvasive peripheral nerve stimulation device programmed to sham mode.
  Arms: Sham neurostimulation
Device: NTX100 Neuromodulation System - Open-Label — Noninvasive peripheral nerve stimulation device programmed to active mode.
  Arms: Open-Label

SUMMARY:
Multi-center, prospective double-blind randomized controlled pivotal study of noninvasive peripheral nerve stimulation (NPNS) with the NTX100 Neuromodulation System for patients with medication-refractory moderate-severe primary RLS

DETAILED DESCRIPTION:
The study consists of a series of two 4-week phases:

Phase 1: Prospective, double-blinded, 1:1 randomized (Active treatment: Sham control)

Phase 2: Prospective, non-randomized, non-blinded, Active treatment

ELIGIBILITY:
Inclusion Criteria:

1. Subject has received a medical diagnosis of primary restless legs syndrome (RLS).
2. Subject is refractory to RLS medication (as defined in section 7.3).
3. Subject has moderate-severe RLS symptoms as defined by a score of 15 or greater points on IRLS (International Restless Legs Syndrome Study Group Rating Scale [12]) over the week prior to study entry.
4. Subject has RLS symptoms 2 or more nights per week during the week prior to study entry as defined by a score of 2, 3, or 4 on IRLS question #7.
5. RLS symptoms are most significant in the subject's lower legs and/or feet.
6. RLS symptoms are most significant at bedtime, after bedtime, and/or in the 2 hours before bedtime.
7. RLS symptoms between 10am and 6pm are not severe.
8. Subject agrees to not change dosage or schedule of any medications that are known to impact RLS symptoms during the study, including RLS medications, antidepressants, sleep medications, or sedative antihistamines.
9. Subject agrees to not make major lifestyle changes during the study including diet, exercise, career, or other changes that would affect bedtime.
10. Subject possesses the necessary equipment, internet/phone accessibility, and communication ability to complete electronic questionnaires and respond to electronic communications and phone calls from the research staff throughout the in-home portion of the study.
11. Subject is ≥ 22 and ≤ 79 years of age when written informed consent is obtained.
12. Subject has signed a valid, Institutional Review Board (IRB)-approved informed consent form, can understand the requirements of the study and instructions for device usage, and can converse in English

Exclusion Criteria:

1. Subject has RLS that is known to be caused by another diagnosed condition (i.e. secondary RLS).
2. Subject is taking an unstable or inconsistent dose or schedule of medication that is likely to impact RLS symptoms, such as antidepressants, sleep medications, or sedative antihistamines or has changed dosage within the past 30 days.
3. Subject has changed dose and schedule of RLS medications within the month prior to study entry or is otherwise on an inconsistent dose or schedule of RLS medications.
4. Subject reports having significant prior experience with neurostimulation devices (including but not limited to transcutaneous electrical nerve stimulation (TENS) devices) or subject has prior experience with neurostimulation devices developed by the study sponsor.
5. Subject was misdiagnosed with RLS, as determined by the investigator (e.g. actual diagnosis of Periodic Limb Movement Disorder (PLMD), arthritis, leg spasms or neuropathy without comorbid RLS).
6. Subject has a sleep disorder other than RLS that interferes with sleep at the present time (except for obstructive sleep apnea that is stably controlled via Continuous Positive Airway Pressure (CPAP)).
7. Subject has active medical device implant anywhere in the body (including but not limited to pacemakers, spinal cord stimulators, deep brain stimulators) or metal implant in the leg.
8. Subject has failed a nerve conduction study prescribed by a physician or has been diagnosed with severe peripheral neuropathy.
9. Subject reports that bedtime is typically outside of 9pm-3am or reports that bedtime regularly varies by more than 4 hours, such as due to shift work.
10. On nights with no RLS symptoms (if any), subject reports typical sleep onset latency of >60min.
11. Subject has been diagnosed with one of the following conditions:

    * Epilepsy or other seizure disorder
    * Current, active or acute or chronic infection other than common cold
    * A malignancy within the past 5 years (not including basal or squamous cell skin cancer)
    * Stage 4-5 chronic kidney disease or renal failure
    * Severe movement disorder symptoms (Parkinson's disease, Huntington's disease, dyskinesia, dystonia)
    * Deep vein thrombosis
    * Multiple sclerosis
12. Subject has moderate or severe cognitive disorder or mental illness.
13. Subject has current diagnosis of iron-deficient anemia or history of iron-deficient anemia within the past year.
14. Subject has known allergy to device materials, electrode gel, polyurethane foam, or lycra (or severe previous reaction to medical adhesives or bandages).
15. Subject has severe edema affecting lower legs.
16. Subject has any of the following at or near the location of device application.

    * Acute injury
    * Cellulitis
    * Open sores
    * Other skin condition
17. Subject is on dialysis or anticipated to start dialysis while participating in the study.
18. During the NTX100 calibration process, which is identical for subjects in the active and sham arms, subject reports not feeling stimulation sensations up to an intensity of 30mA or finds stimulation intensities less than 15 milliamperes (mA) to be uncomfortable or distracting.
19. Subject has received another investigational device or drug within 30 days before study entry, is planning to receive another investigational device or drug during the study, or is planning to change RLS medications during the study.
20. Subject has undergone a major surgery (excluding dental work) in the 30 days prior to study entry.
21. Subject is unable or unwilling to comply with study requirements.
22. Subject is pregnant or trying to become pregnant.
23. Subject has a medical condition not listed above that may affect validity of the study as determined by the investigator.
24. Subject has a medical condition not listed above that may put the subject at risk as determined by the investigator

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Charlesworth, PhD, Study Director — Noctrix Health, Inc.
Locations (7):
- United States (7):
  - California Center for Sleep Disorders, San Leandro, California
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Neurotrials Research, Atlanta, Georgia
  - Clayton Sleep Institute, St Louis, Missouri
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas

REFERENCES:
- [Derived] Bogan RK, Roy A, Kram J, Ojile J, Rosenberg R, Hudson JD, Scheuller HS, Winkelman JW, Charlesworth JD. Efficacy and safety of tonic motor activation (TOMAC) for medication-refractory restless legs syndrome: a randomized clinical trial. Sleep. 2023 Oct 11;46(10):zsad190. doi: 10.1093/sleep/zsad190. PMID 37458698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects must have received a medical diagnosis of primary restless legs syndrome (RLS), have moderate-severe RLS and be refractory to RLS medication.
Groups:
- TOMAC Group: Stage 1 (4 weeks): Double-blind, Noninvasive peripheral nerve stimulation device programmed to deliver active stimulation
  Stage 2 (4 weeks): Open-label, noninvasive peripheral nerve stimulation device programmed to active mode.
- Sham Control Group: Stage 1 (4 weeks): Double-blind, Noninvasive peripheral nerve stimulation device programmed to deliver SHAM stimulation
  Stage 2 (4 weeks): Open-label, noninvasive peripheral nerve stimulation device programmed to active mode.
Period: Overall Study
Arm/Group | TOMAC Group | Sham Control Group
Started | 68 | 65
Completed | 65 | 62
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- TOMAC Group: Noninvasive peripheral nerve stimulation device programmed to deliver active stimulation - Phase 1
  NTX100 Neuromodulation System - Active: Noninvasive peripheral nerve stimulation device programmed to active mode.
- Sham Control Group: Noninvasive peripheral nerve stimulation device programmed to deliver non-therapeutic (sham) stimulation - Phase 1
  NTX100 Neuromodulation System - Sham: Noninvasive peripheral nerve stimulation device programmed to sham mode.
- Total: Total of all reporting groups
Arm/Group | TOMAC Group | Sham Control Group | Total
Number analyzed (Participants) | 68 | 65 | 133
Age, Customized [Mean (Standard Deviation); unit: years] | 56.3 (10.96) | 58.6 (11.81) | 57.46 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 29 | 24 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 64 | 61 | 125
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 64 | 65 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
IRLS Total Score at Baseline [Mean (Standard Deviation); unit: Units on a scale] — International Restless Legs Score (IRLS) is a participant-rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe.
  Units on a scale | 25.2 (5.3) | 25.4 (5.3) | 25.3 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects for Which the Clinician Reported "Much Improved" or "Very Much Improved" on the Clinical Global Impressions-Improvement (CGI-I) Scale for TOMAC Compared to Sham
Description: Responder rate is defined as the proportion of responses of "Much Improved" or "Very Much Improved" relative to baseline on the investigator-rated 7-point CGI-I scale.
Time Frame: Week 4
Population: Primary Efficacy Endpoint (CGI-I Responder Rate at Week 4) - (ITT Population)
Measure: Count of Participants; unit: Participants
Arm/Group | TOMAC Group | Sham Control Group
Number analyzed (Participants) | 68 | 65
Participants | 29 | 10

2. Secondary Outcome: Responder Rate on Patient Global Impressions-Improvement (PGI-I) Scale
Description: Responder rate is defined as the proportion of responses of "Much Improved" or "Very Much Improved" relative to baseline on the participant-rated 7-point PGI-I scale.
Time Frame: Week 4
Population: Key Secondary Efficacy Endpoints (ITT Population)
Measure: Count of Participants; unit: Participants
Arm/Group | TOMAC Group | Sham Control Group
Number analyzed (Participants) | 68 | 65
Participants | 33 | 12

3. Secondary Outcome: Mean Change From Baseline in International Restless Legs Syndrome Study Group Rating Scale (IRLS) Score
Description: IRLS is a participant-rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe.
Time Frame: Week 4
Population: Key Secondary Efficacy Endpoints (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- TOMAC Group; Sham Control Group: Stage 1 (4 weeks): Double-blind, Noninvasive peripheral nerve stimulation device programmed to deliver SHAM stimulation
  Stage 2 (4 weeks): Open-label, noninvasive peripheral nerve stimulation device programmed to active mode.
Arm/Group | TOMAC Group | Sham Control Group
Number analyzed (Participants) | 68 | 65
score on a scale | -7.2 (6.2) | -3.8 (5.9)

4. Secondary Outcome: Mean Change From Baseline in Medical Outcomes Study Sleep Problems Index II (MOS-II) Score
Description: MOS-II is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality. The MOS-I (6-items) and MOS-II (9-items) are the two validated subscales of the 12-item MOS Sleep Scale. Both are scored from 0 to 100, where 100 corresponds to the worst possible sleep problems and 0 corresponds to no sleep problems. See https://labs.dgsom.ucla.edu/hays/files/view/docs/surveys/sleep/sleepman-112603.pdf for more information.
Time Frame: Week 4
Population: Key Secondary Efficacy Endpoints (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOMAC Group | Sham Control Group
Number analyzed (Participants) | 68 | 65
score on a scale | -13.7 (14.9) | -4.0 (14.8)

5. Secondary Outcome: Mean Change From Baseline in Medical Outcomes Study Sleep Problems Index I (MOS-I) Score
Description: MOS-I is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality. The MOS-I (6-items) and MOS-II (9-items) are the two validated subscales of the 12-item MOS Sleep Scale. Both are scored from 0 to 100, where 100 corresponds to the worst possible sleep problems and 0 corresponds to no sleep problems. See https://labs.dgsom.ucla.edu/hays/files/view/docs/surveys/sleep/sleepman-112603.pdf for more information.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOMAC Group | Sham Control Group
Number analyzed (Participants) | 68 | 65
score on a scale | -11.8 (14.7) | -2.8 (14.9)

6. Secondary Outcome: Mean Clinical Global Impressions-Improvement (CGI-I) Scale Rating
Description: Mean rating on the investigator-rated 7-point Likert CGI-I scale, where lower scores indicate improvement. Possible choices (followed by scale value) are: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very Much Worse (7).
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TOMAC Group | Sham Control Group
Number analyzed (Participants) | 68 | 65
score on a scale | 2.6 (1.1) | 3.5 (0.9)

7. Secondary Outcome: Score for Question #7 of the International Restless Legs Syndrome Study Group Rating Scale (IRLS)
Description: Question #7 of the IRLS assesses the participant-rated frequency (days/week) of RLS symptoms on a scale from 0 to 4, where lower scores indicate less frequent symptoms
Time Frame: Week 8
Population: Key Secondary Efficacy Endpoints (ITT Population)
Measure: Mean (Standard Deviation); unit: Days per Week
Arm/Group | TOMAC Group | Sham Control Group
Number analyzed (Participants) | 68 | 65
Days per Week | -0.9 (1.07) | -0.6 (1.2)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Descriptive analyses of adverse events for both study arms, classified and tabulated by seriousness, relationship to the device, and severity.
Groups:
- TOMAC Group: Treatment group
- Sham Control Group: Control group
Arm/Group | TOMAC Group | Sham Control Group
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/65
Other Adverse Events (participants affected / at risk) | 28/68 | 23/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOMAC Group (N=68) | Sham Control Group (N=65)
Administration site discomfort (Skin and subcutaneous tissue disorders) | 22 (22) | 16 (16)
Administration site irritation (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04874155/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT04874155/SAP_001.pdf